CLINICAL TRIAL: NCT01700907
Title: Optimization of Desflurane in Elderly Patients Compared With Sevoflurane: A Pilot Study
Brief Title: Optimization of Desflurane in Elderly Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sapporo Medical University (Other)
Responsible Party: Principal Investigator, Michiaki Yamakage, Optimization of Desflurane in Elderly Patients Compared with Sevoflurane: A Pilot Study, Sapporo Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DES-40-POCD
Record Dates: First submitted 2012-09-30; First posted 2012-10-04 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative cognitive dysfunction; elderly patients; long surgery
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group DES (Active Comparator): The patients in this arm will be given the general anesthesia with desflurane and be used the Aysis as the anesthetic machine.
  Interventions: Drug: Desflurane
- group SEVO (Active Comparator): The patients in this arm will be given the general anesthesia with sevoflurane and be used the Aysis as the anesthetic machine.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane — The patients in this arm will be given the general anesthesia with desflurane and be used the Aysis as the anesthetic machine.
  Other Names: (2RS)-2-(Difluoromethoxy)-1,1,1,2-tetrafluoroethane
  Arms: group DES
Drug: Sevoflurane — The patients in this arm will be given the general anesthesia with sevoflurane and be used the Aysis as the anesthetic machine.
  Other Names: 1,1,1,3,3,3-Hexafluoro-2-(fluoromethoxy)propane
  Arms: group SEVO

SUMMARY:
Various issues had been pointed out when undergoing the anesthesia for elderly patients with sevoflurane, such as delayed emergence, post-operative trouble with swallowing.

Desflurane, which has a lower blood/gas partition coefficient, is expected to contribute the better emergence, along with the recent progress on optimization of delivered amount of anesthesia.

The purpose of this study is to compare the time to emergence in long elderly patient cases with desflurane or sevoflurane, with the recently developed drug-delivery optimization system "Aisys®" (GE Healthcare Japan).

DETAILED DESCRIPTION:
The objectives of this study is to compare the time to emergence and quality of recovery in long elderly patient cases with desflurane or sevoflurane, with the recently developed drug-delivery optimization system "Aisys®" (GE Healthcare Japan).

Inclusion Criteria:

- Elderly patients (>= 65 yr-old), long operation (> 4hours), abdominal surgery patients

Exclusion Criteria:

- Liver dysfunction, Renal dysfunction, preoperative dementia Neurosurgery patients, Cardiac surgery patients, obese patients(BMI>35)

ELIGIBILITY:
Inclusion Criteria:

- Elderly patients (>= 65 yr-old), long operation (> 4hours), abdominal surgery patients

Exclusion Criteria:

- Liver dysfunction, Renal dysfunction, preoperative dementia Neurosurgery patients, Cardiac surgery patients, obese patients(BMI>35)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michiaki Yamakage, M.D.,PhD, Principal Investigator — Sapporo Medical University, School of Medicine
Locations (1):
- Sapporo Medical University, School of Medicine, Sappro, Hokkaido, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty patients who were scheduled to undergo general anesthesia in Sapporo Medical University Hospital were enrolled in this study.
Pre-assignment Details: Inclusion criteria were shown as follows: Elderly patients (>= 65 yr-old), long operation (> 4hours), abdominal surgery patients.
  Exclusion criteria were shown as follows: Liver dysfunction, Renal dysfunction, preoperative dementia Neurosurgery patients, Cardiac surgery patients, obese patients (BMI>35)
Period: Overall Study
Arm/Group | Group DES | Group SEVO
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group DES | Group SEVO | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (6.0) | 74.1 (6.5) | 74.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Japan | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Time From the End of Anesthesia to Extubation
Description: When surgery ends, the fresh gas flow rate will be increased to 6L/min (100% oxygen). Patients will be asked to open eyes by touching the shoulder, calling the name every 15 seconds. Patients will be applied stimulus every 15 seconds until following commands. Extubation will be performed when the patient is judged to be awake and spontaneous breathing recovery substantially.
Time Frame: Within 60 minutes after the end of anesthesia
Population: This is a pilot study.
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Group DES | Group SEVO
Number analyzed (Participants) | 10 | 10
second | 329.0 [296.2 to 453.0] | 636.0 [613.5 to 918.8]

2. Secondary Outcome: The Time From the End of Anesthesia to Eye Opening
Description: as for outcome 1
Time Frame: Within 60 minutes after the end of anesthesia
Population: This is a pilot study.
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Group DES | Group SEVO
Number analyzed (Participants) | 10 | 10
second | 176.5 [166.0 to 317.0] | 315.0 [277.2 to 404.8]

3. Secondary Outcome: The Time From the End of Anesthesia to Following Commands
Description: as for outcome 1
Time Frame: Within 60 minutes after the end of anesthesia
Population: This is a pilot study.
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Group DES | Group SEVO
Number analyzed (Participants) | 10 | 10
second | 246.5 [169.1 to 357.3] | 424.0 [352.3 to 553.0]

4. Secondary Outcome: Cognitive Function
Description: Cognitive function will be measured by MMSE (Mini-Mental State Examination) at 24hrs pre and postoperatively. Total MMSE score is recorded by interview ranging from 0 (minimum) to 30 (maximum). MMSE score is consisted on 11 subscales, and total MMSE score is simply summation of all the subscale scores. Maximum MMSE score indicates that the patient is excellent for cognitive function. MMSE score under 26 indicated the cognitive dysfunction.
Time Frame: 24 hrs pre and postoperatively
Population: This is a pilot study
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Group DES | Group SEVO
Number analyzed (Participants) | 10 | 10
Scores on a scale
  pre-operation | 28.0 [27.0 to 29.0] | 28.0 [27.5 to 29.0]
  post-operation | 29.5 [28.0 to 30.0] | 29.0 [28.3 to 30.0]

5. Secondary Outcome: The Incidence of Postoperative Delirium
Description: The incidence of post operative delirium will be measured by Confusion Assessment Method (CAM) at baseline, 15mins, 3hrs, 6hrs, 12hrs, 24hrs, 48hrs postoperatively.
Time Frame: from 15 minutes to 48 hrs postoperatively
Population: This is a pilot study.
Measure: Number; unit: participants
Arm/Group | Group DES | Group SEVO
Number analyzed (Participants) | 10 | 10
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: The adverse event will be evaluated at 24 h after surgery by interviewing.
Description: The adverse event is defined as follows: postoperative death, re-operation, hypotension (systolic blood pressure under 80 mmHg), and delirium at 24 h after surgery. If the adverse event occur and recover until 24 h after surgery, the adverse event is not counted. Other adverse event is not assessed.
Arm/Group | Group DES | Group SEVO
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No